CLINICAL TRIAL: NCT04202445
Title: TreatMent of ActInic KerAtosis Lesions : pharmacoepiDemiological Study of the Impact in Real Life of ingenOl Mebutate Gel (Picato®) on Patients Satisfaction
Acronym: MIKADO
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-PICATO-1087
Record Dates: First submitted 2015-09-15; First posted 2019-12-17 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2019-12

CONDITIONS: Actinic Keratosis
Keywords: Actinic keratosis; Field treatment; Ingenol mebutate; Picato; Mikado
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ingenol mebutate — Topical field treatment as prescribed by dermatologist
  Other Names: Picato

SUMMARY:
This is an observational longitudinal study, prospective, multicenter, performed in metropolitan France, on a representative sample of dermatologists.

Data will be collected by physicians during 2 or 3 visits (according to their usual practice), from the patient file, questioning and clinical examination performed during these visits.

Data about the patient's perception (satisfaction, perception of local skin reactions, quality of life) will be collected directly by the patient using self-administered questionnaires at inclusion visit, day 7 and 2 months later.

DETAILED DESCRIPTION:
Actinic keratosis (AKs) are common skin diseases affecting areas previously overexposed to the sun (in particular face, nape of the neck, hands). They affect mainly elderly people (mean age: 74 years old, with 97% who are over 50 years old) and preferably men (60%). In Europe, prevalence of AK in the adult population over 40 years is estimated to be between 6% and 25%.

Subjects at risk are light-skinned people (phototype I and II according to Fitzpatrick scale) with high cumulative sun exposure or phototherapy. Over 80% of patients have a light phototype and 37% of patients with AK have an outside professional activity.

Diagnosis of AK is usually clinical, during skin examination which is recommended for any physician's visit. There are often multiple lesions, some of which, in the absence of effective treatment, can progress to squamous cell carcinoma (0.025% to 20% per year/lesion).

Although the evolution rate of AKs to carcinoma remains low and disappearance or sole persistence of the lesion is possible, their evolution is unpredictable, and it is therefore recommended to monitor and treat the AKs.

Treatment options include cryotherapy, topical treatments, photodynamic therapy, vaporization of lesions by CO2 laser or electrocoagulation and curretage.

When there are few AK lesions, which are localized and with superficial forms, cryotherapy is the reference treatment (it is widely used by dermatologists, as it is simple, fast and does not require special equipment), whereas topical treatment (5-FU, imiquimod, diclofenac) is recommended in case of multiple keratosis or lesions on a larger area of the skin. The disadvantage of cryotherapy and photodynamic therapy is that these techniques can be painful and lead to depigmentation or scarring. Topical treatments which are available (imiquimod, 5-FU, diclofenac) may induce severe inflammatory reactions sometimes responsible for premature termination and thus ineffective.

Combined with their length (4 to 16 weeks), the complexity of current topical regimens would be the cause of poor compliance.

So, all dermatologists agree with the need to shorten duration of treatment and reduce the number of applications. Ingenol mebutate gel (Picato®), used in very short 2-3 days cycle, with one application per day, meets this need.

Development of ingenol mebutate gel included 4 pivotal phase III trials, evaluating its efficacy and safety. The results of these studies have established satisfactory efficacy and safety for Picato® with, on one hand, proven efficacy after two months for face, scalp, trunk and extremities and, on the other hand, transient local skin reactions (erythema, flaking/scaling, crusting,swelling,...), which appear early, peak in intensity after the end of treatment (day 3 or day 4) and disappear without sequelae within 2-4 weeks after application of the gel. At day 57, mean patient global satisfaction scores, either assessed with TSQM or Skindex-16, were statistically higher in the ingenol mebutate gel group than in the vehicle group. In a long term follow up study, ingenol mebutate produced clinically relevant sustained clearance and long-term lesion reduction.

These characteristics are a potentially important advantage for treatment compliance as well as for patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old, seen by the dermatologist during a consultation, whether actinic keratosis is the reason for consultation or not.
* Patient with AK lesions and for whom the dermatologist decided to initiate a treatment with Picato®* 150 or Picato®* 500
* Patient informed and accepting the automatic processing of medical data * To respect the physicians' independence, this study is conducted among patients for whom the decision of therapeutic care is not related to their inclusion.

Exclusion Criteria:

* Patient with a contraindication to treatment with Picato®.
* Patient unable to read and/or to understand a self-administered questionnaire.
* Patient already included in the study.
* Patient participating or having participated in the previous month in a clinical trial in dermatology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with actinic keratosis planned to receive treatment with ingenol mebutate at the discretion of the dermatologist
Sampling Method: Non-Probability Sample
Enrollment: 1218 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Treatment Satisfaction Questionnaire of Medication (TSQM-9) | 2 months after end of treatment
  The TSQM-9 scale is a 7-item instrument to be completed by patients. The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domaine.

SECONDARY OUTCOMES:
Dermatology Life Quality Index - DLQI | Baseline and 2 months after end of treatment
  Dermatology Life Quality Index is an index based on a series of 10 questions, each scored on a verbal rating scale with 2 to 4 answer categories, and except for three questions the option to state that the question is not relevant. The DLQI score is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
Real-life efficacy of Picato | Between Day 1 after the treatment application and 12 months (maximum 2 follow-up visits after the inclusion)
  Efficacy assessed using the following scale filled out by the physician:
  - How do you assess the treatment efficacy : 1-Excellent / 2-Good / 3-Mild / 4-Bad / 5-NA

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Moumane, MD, Study Chair — LEO Pharma

REFERENCES:
- [Background] Frost CA, Green AC. Epidemiology of solar keratoses. Br J Dermatol. 1994 Oct;131(4):455-64. doi: 10.1111/j.1365-2133.1994.tb08544.x. PMID 7947197
- [Background] Memon AA, Tomenson JA, Bothwell J, Friedmann PS. Prevalence of solar damage and actinic keratosis in a Merseyside population. Br J Dermatol. 2000 Jun;142(6):1154-9. doi: 10.1046/j.1365-2133.2000.03541.x. PMID 10848739
- [Background] Quaedvlieg PJ, Tirsi E, Thissen MR, Krekels GA. Actinic keratosis: how to differentiate the good from the bad ones? Eur J Dermatol. 2006 Jul-Aug;16(4):335-9. PMID 16935787
- [Background] Dinehart SM. The treatment of actinic keratoses. J Am Acad Dermatol. 2000 Jan;42(1 Pt 2):25-8. doi: 10.1067/mjd.2000.103338. PMID 10607354
- [Background] French Society of Dermatology. [Guidelines for the diagnosis and treatment of cutaneous squamous cell carcinoma and precursor lesions. Arguments - May 2009]. Ann Dermatol Venereol. 2009 Sep;136 Suppl 5:S189-242. No abstract available. French. PMID 19795558
- [Background] Thai KE, Fergin P, Freeman M, Vinciullo C, Francis D, Spelman L, Murrell D, Anderson C, Weightman W, Reid C, Watson A, Foley P. A prospective study of the use of cryosurgery for the treatment of actinic keratoses. Int J Dermatol. 2004 Sep;43(9):687-92. doi: 10.1111/j.1365-4632.2004.02056.x. PMID 15357755
- [Background] Burge SM, Bristol M, Millard PR, Dawber RP. Pigment changes in human skin after cryotherapy. Cryobiology. 1986 Oct;23(5):422-32. doi: 10.1016/0011-2240(86)90027-1. PMID 3769517
- [Background] Zouboulis CC. Cryosurgery in dermatology. Eur J Dermatol. 1998 Oct-Nov;8(7):466-74. PMID 9854156
- [Background] Fu W, Cockerell CJ. The actinic (solar) keratosis: a 21st-century perspective. Arch Dermatol. 2003 Jan;139(1):66-70. doi: 10.1001/archderm.139.1.66. No abstract available. PMID 12533168
- [Background] Lebwohl M, Swanson N, Anderson LL, Melgaard A, Xu Z, Berman B. Ingenol mebutate gel for actinic keratosis. N Engl J Med. 2012 Mar 15;366(11):1010-9. doi: 10.1056/NEJMoa1111170. PMID 22417254
- [Background] Anderson L, Schmieder GJ, Werschler WP, Tschen EH, Ling MR, Stough DB, Katsamas J. Randomized, double-blind, double-dummy, vehicle-controlled study of ingenol mebutate gel 0.025% and 0.05% for actinic keratosis. J Am Acad Dermatol. 2009 Jun;60(6):934-43. doi: 10.1016/j.jaad.2009.01.008. PMID 19467365
- [Background] Berman B. New developments in the treatment of actinic keratosis: focus on ingenol mebutate gel. Clin Cosmet Investig Dermatol. 2012;5:111-22. doi: 10.2147/CCID.S28905. Epub 2012 Aug 24. PMID 22956883